CLINICAL TRIAL: NCT01771900
Title: Heart Failure Exercise and Resistance Training CAMP
Brief Title: Heart Failure Exercise And Resistance Training Camp (HEART Camp)
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0050-05-FB; 1R15NR009215-01 (NIH)
Record Dates: First submitted 2012-06-15; First posted 2013-01-18 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: heart failure; exercise; adherence to exercise
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart Camp Group (Experimental): In Week 1, 2, and 3 subjects will attend the HEART CAMP. Subjects will set specific exercise goals. Subjects will be taught how to record exercise data on the computer at the exercise facility. Specific activities will teach subjects aerobic and resistance training exercises and build self-efficacy to exercise. During the period from month 3 to the end of study subjects will continue the training program independently and no formal sessions will be scheduled.
  Interventions: Behavioral: Heart Camp Group
- Attention Control Group (Experimental): Subjects will receive a 60 minute group session led by a specifically designated control group intervention nurse. Phone calls will be placed to the subject if they miss a Friday group session and attendance to meetings will be encouraged.
  Interventions: Behavioral: Attention Control Group

INTERVENTIONS:
Behavioral: Heart Camp Group — In Week 1, 2, and 3 subjects will attend the HEART CAMP. Subjects will set specific exercise goals. Subjects will be taught how to record exercise data on the computer at the exercise facility. Specific activities will teach subjects aerobic and resistance training exercises and build self-efficacy to exercise. During the period from month 3 to the end of study subjects will continue the training program independently and no formal sessions will be scheduled.
  Arms: Heart Camp Group
Behavioral: Attention Control Group — Subjects will receive a 60 minute group session led by a specifically designated control group intervention nurse. Phone calls will be placed to the subject if they miss a Friday group session and attendance to meetings will be encouraged.
  Arms: Attention Control Group

SUMMARY:
The purpose of this feasibility study was to obtain pilot data, as the basis for a future, larger investigation, testing the impact of an innovative training camp intervention called HEART CAMP (Heart failure Exercise And Resistance Training CAMP) to teach HF patients how to exercise and self-manage exercise behavior over time. The study assessed the feasibility and adequacy of the intervention, the data collection plan, and the reliability and sensitivity of the outcome measures. The 6-month intervention was based on a training camp model to teach HF patients how to exercise in a fun, group-oriented atmosphere. Subjects interacted and exercised in small groups with an exercise physiologist and nurse to guide activities. The dosage of the intervention (frequency and amount of direct guidance from the exercise physiologist and nurse) decreased over the 6 months in order to increase subject's independence and promote long-term adherence to exercise. The intervention incorporated use of computerized data files to monitor exercise behavior, compare exercise performance to individualized goals and provide feedback as strategies to foster adherence and self-management of exercise behavior.

DETAILED DESCRIPTION:
This study uses an experimental repeated measures design with randomized comparison of the HEART CAMP intervention group and the attention control group. The purpose of this feasibility study is to obtain pilot data, as the basis for a future, larger investigation, testing the impact of an innovative 24-week (6-month) training camp intervention (HEART CAMP). HEART CAMP is designed to teach heart failure (HF) patients how to exercise (aerobic and resistance) and self-manage exercise behavior over time. Patients receiving care at the BryanLGH Heart Institute heart failure clinic will be eligible for the study.

The HEART CAMP intervention is a multi-component intervention derived from Bandura's cognitive behavioral theory and consists of specific strategies to build self-efficacy for exercise. The subject, under the guidance of an exercise physiologist and nurse, will be taught how to exercise (aerobic and resistance). A baseline cardiopulmonary exercise test will be completed on all subjects. The first three weeks of HEART CAMP will be held in a hospital based cardiac rehabilitation department where subjects will be electrocardiographically monitored during the five-day per week training sessions. Training sessions will be delivered in cohort groups of eight subjects and will focus on exercise, self-evaluation of response to exercise, and group debriefing sessions for problem solving and relapse management. Weeks 4 through 12 subjects will complete three aerobic exercise sessions in the cardiac rehabilitation maintenance facility and two resistive training sessions at home with the exercise physiologist and nurse monitoring subject response and delivering group debriefing sessions each week. Weeks 12 through 24 subjects exercise independently with the exercise physiologist and nurse monitoring subject exercise data and available as needed.

The attention control group will receive weekly cohort group education sessions during the first 3 months similar to the intervention groups' participation in weekly group sessions. One week an educational topic will be presented and the subsequent week the cohort group of eight subjects will discuss the topic. Six topics will be presented including: Eating Fruits, Vegetables, and Grains; Shopping Wisely; Cooking Healthy; Time Management; Communicating Assertively; and Learning to Relax.

Outcome measures will be completed at baseline, 3 weeks, 3 and 6 months (end of study) for both groups. Primary outcomes are estimated energy expenditure, self-efficacy to exercise, and adherence to exercise. Secondary outcomes are symptoms, biomarker (BNP), physical and psychological functioning and quality of life

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or greater
* Oriented to person, place, time
* Able to speak and read English
* Resting left ventricular ejection fraction of 40% of less
* Optimum stable medical therapy for past 30 days

Exclusion Criteria:

* Clinical evidence of decompensated HF
* Unstable angina pectoris
* Myocardial infarction, coronary artery bypass surgery or biventricular pacemaker less than 3 months ago
* Orthopedic or neuromuscular disorders preventing participation in exercise and strength/resistance training
* Participation in 3 times per week aerobic exercise during the past 12 months.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-04-01 (Actual); Primary Completion 2007-12-26 (Actual); Study Completion 2007-12-26 (Actual)

PRIMARY OUTCOMES:
Adherence to Exercise | Baseline to 3 months
  Change in adherence to exercise as recorded in digital diary
Change in Self-efficacy to exercise | Baseline to three months
  Measured with the Cardiac Exercise Self-Efficacy Instrument
Change in Estimated energy expenditure | Baseline to three months
  Measured with the RT3 Accelerometer

SECONDARY OUTCOMES:
Change in Symptoms | Baseline to three months
  Measured with the Dyspnea-Fatigue Index
Change in Biomarkers | Baseline to three months
  BNP is an effective, reliable and powerful cardiac biomarker for early diagnosis heart failure (HF). BNP are small proteins produced in left-ventricular myocardium, when there is an excess of fluids that causes myocardial stretch. The normal concentration of BNP in blood is 35pg/mL.
Change in Physical and psychological functioning | Baseline to three months
  Measured by the MOS SF-36
Heart failure symptoms impact on physical and social function and quality of life | Baseline to three months
  Measured with the Kansas City Cardiomyopathy Questionnaire, a self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bunny Pozehl, PhD, APRN-NP, Principal Investigator — University of Nebraska
Locations (1):
- BryanLGH Heart Institute, Lincoln, Nebraska, United States

REFERENCES:
- [Result] Pozehl B, Duncan K, Hertzog M, Norman JF. Heart Failure Exercise And Training Camp: effects of a multicomponent exercise training intervention in patients with heart failure. Heart Lung. 2010 Nov-Dec;39(6 Suppl):S1-13. doi: 10.1016/j.hrtlng.2010.04.008. Epub 2010 Jul 3. PMID 20598373
- [Result] Norman JF, Pozehl BJ, Duncan KA, Hertzog MA, Elokda AS, Krueger SK. Relationship of resting B-type natriuretic peptide level to cardiac work and total physical work capacity in heart failure patients. J Cardiopulm Rehabil Prev. 2009 Sep-Oct;29(5):310-3. doi: 10.1097/HCR.0b013e3181ac7bcb. PMID 19561522
- [Result] Duncan K, Pozehl B, Norman JF, Hertzog M. A self-directed adherence management program for patients with heart failure completing combined aerobic and resistance exercise training. Appl Nurs Res. 2011 Nov;24(4):207-14. doi: 10.1016/j.apnr.2009.08.003. Epub 2009 Oct 15. PMID 22099469